CLINICAL TRIAL: NCT05891561
Title: Short-course Trastuzumab, Pertuzumab Combined with Taxanes in the Adjuvant Treatment of Early Human Epidermal Growth Factor Receptor 2-positive Breast Cancer: an Open-label, Single-arm Study
Brief Title: Short-course Trastuzumab, Pertuzumab with Taxanes in the Adjuvant Treatment of Early HER2-positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC-THP4
Record Dates: First submitted 2023-05-21; First posted 2023-06-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; pertuzumab; her2; adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pertuzumab (Experimental): 4 cycles of taxane, Pertuzumab, Trastuzumab
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — 4 cycles of taxane, pertuzumab, trastuzumab

SUMMARY:
The investigators plan to carry out a phase II, open-label, single-arm clinical study of short-course trastuzumab, pertuzumab combined with taxanes in the adjuvant treatment of early HER2-positive breast cancer, to explore whether 4 courses of dual HER2 blockade combined with taxanes can lead to a similar prognosis with current standard treatment, which is one-year trastuzumab monotherapy combined with chemotherapy, while reducing the adverse reactions of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed unilateral primary invasive breast cancer patient with pT1, pN0, and M0 disease
* HER2-positive, ie. immunohistochemistry [IHC] 3+ or IHC 2+ and fluorescence in situ hybridisation [FISH]-positive according to ASCO/CAP 2018 guidelines
* complete clinical pathological information
* Eastern Cooperative oncology Group [ECOG] 0-1
* Currently not pregnant or breast-feeding
* Fine organ function
* Have good compliance with planned treatment, understand the study process and sign a written informed consent

Exclusion Criteria:

* Bilateral or metastatic breast cancer
* Receiving neoadjuvant treatment
* Other malignancies within 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer
* Severe systemic infections or other serious illnesses
* HIV infection, active hepatitis B or C infection
* Known allergy to or intolerance to a therapeutic drug or its excipients
* Prior history of chemotherapy, endocrine therapy, biotherapy, or radiation therapy for any reason
* Enrollment of another investigational study within 4 weeks prior to initial administration of the investigational treatment
* Receiving live vaccine within 30 days prior to initial administration of the investigational treatment
* History of mental illness or drug abuse that may affect compliance with the trial requirements
* The researchers determine that the patients were not suitable for the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival [DFS] | 3 year
  Time from surgery to first proven loco-regional recurrence, distant recurrence, second non-breast malignancy, or death from any cause

SECONDARY OUTCOMES:
Overall survival [OS] | 3 year
  Time from surgery to death from any cause
Distant disease-free survival [DDFS] | 3 year
  Time from surgery to first proven distant recurrence, second non-breast malignancy, or death from any cause
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No